CLINICAL TRIAL: NCT04567823
Title: Human Intervention Study for Validating Nutrient Bioavailability From Microalgae
Brief Title: Nutrient Bioavailability From Microalgae
Acronym: NovAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, Study leader, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H10_20
Record Dates: First submitted 2020-09-15; First posted 2020-09-29 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-09

CONDITIONS: Nutrient Deficiency
Keywords: microalgae; omega-3 fatty acids; vitamins; minerals; trace elements

STUDY DESIGN:
Intervention Model Description: parallel design
Who Masked: Participant, Care Provider, Investigator
Masking Description: It is not visible whether the smoothie is fortified with microalgae or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Microalgae I (Experimental): Smoothie (enriched with Chlorella pyrenoidosa) and standardised background diet (defined menu plans)
  Interventions: Dietary Supplement: Smoothie with microalgae
- Microalgae II (Experimental): Smoothie (enriched with Nannochloropsis salina) and standardised background diet (defined menu plans)
  Interventions: Dietary Supplement: Smoothie with microalgae
- Smoothie (Placebo Comparator): Smoothie (without microalgae) and standardised background diet (defined menu plans)
  Interventions: Dietary Supplement: Smoothie with microalgae
- Control (No Intervention): no intervention (no smoothie, no menu plans)

INTERVENTIONS:
Dietary Supplement: Smoothie with microalgae — Smoothie with microalgae I: Chlorella pyrenoidosa, Smoothie with microalgae II: Nannochloropsis salina, Smoothie without microalgae
  Arms: Microalgae I; Microalgae II; Smoothie

SUMMARY:
The intervention study is designed to evaluate nutrient bioavailability and physiological impact of two selected microalgae species of interest in a randomized study in humans. The controlled study in parallel design will be conducted with healthy males and females between 20 and 35 years.

DETAILED DESCRIPTION:
The microalgae are selected depending on their contents of long-chain omega-3 fatty acids, e.g. eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), high-quality protein (focus: essential amino acids), dietary fibers but also vitamin D pre-cursors and further vitamins, minerals and trace elements.The nutrient bioavailability is evaluated in a controlled, randomized, double-blind study in parallel design. The intervention products (smoothie enriched with Chlorella pyrenoidosa, Nannochloropsis salina) are consumed daily over 14 days. In addition, the background diet is standardised by provision of defined menu plans ensuring an optimal energy and nutrient intake. The control group I receive no intervention products and no menu plans and control group II receive a smoothie without microalage and defined menu plans.

A sup-group of five participants per group consume a test meal after the fasting blood sampling on the first study day. This is followed by a postprandial blood sampling after 30, 60, 90, 120 and 180 minutes.

The NovAL study is conducted to evaluate the bioavailability of nutrients such as omega-3 LC-PUFA, vitamin D, vitamin B12, further vitamins, amino acids, minerals, and trace elements from the selected microalgae species. Therefore, the concentration of these valuable nutrients and relevant markers of their status in humans (e.g. vitamin B12 status: holo-transcobalamin, methylmalonic acid, homocysteine; iron status: ferritin, transferrin, transferrin saturation) are analysed in the human biofluids (serum/plasma, erythrocytes, 24 h urine) before and after defined consumption of the selected microalgae species over 14 days. Besides the comprehensive analysis of the nutrient status in humans, cardiovascular risk factors and risk factors for diabetes mellitus type II are analysed. Thus, the NovAL study allows the assessment of i) the nutrient bioavailability from the selected microalgae species but also ii) their contribution on nutrient supply and prevention of non-communicable diseases such as cardiovascular diseases or diabetes mellitus type.

ELIGIBILITY:
Inclusion Criteria:

* females and males
* BMI < 30 kg/m2
* subjects must be able and willing to give written informed consent, and to comply with study procedures
* participants following a traditional Western diet composed of dairy products, sausage, meat, fast foods, chocolate and snacks, cereals, vegetables, and fruits (PAL: 1.6)
* precondition: Stable eating habits of at least one years before enrolment
* subjects must have adequate fluency in the German language to complete the questionnaires and understand the nutritional recommendations

Exclusion Criteria:

* subjects with any acute or chronic disease (CVD, tumor, infection, other), gastrointestinal diseases, diabetes mellitus (type I and II), chronic renal disease, diseases of the parathyroid, diseases necessitating regular phlebotomies other chronic diseases which could affect the results of the present study
* use of prescription medicine which could affect results of the study, including systemic glucocorticoids
* intake of lipid-lowering drugs, diabetes medication, hormone replacement therapy
* estimated glomerular filtration (eGFR) rate < 60 ml/min
* weight loss (≤ 3 kg) or weight gain (≥ 3 kg) during the last three months before study begin
* pregnancy or lactation
* transfusion of blood in the last three months before blood sample taking
* use of dietary supplements incl. multivitamins, fish oil capsules, minerals, and trace elements (three months before and during the entire study period)
* vegetarians, vegans, food allergies
* dependency on alcohol or drugs
* elite athletes (>10 hours of strenuous physical activity per week)
* simultaneous participation in other clinical studies
* inability (physically or psychologically) to comply with the procedures required by the protocol

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
EPA concentration in plasma lipids | change from baseline after 2 weeks
  concentration of eicosapentaenoic acid (EPA) in % fatty acid methyl esthers (FAME) in plasma lipids

SECONDARY OUTCOMES:
blood lipids | change from baseline after 2 weeks
  total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides in mmol/l
anthropometric data | change from baseline after 2 weeks
  body water, body fat, lean body mass, extracellular mass (ECM), body cell mass (BCM) in %
body mass index | change from baseline after 2 weeks
  body mass index (kg/m2)
blood pressure | change from baseline after 2 weeks
  systolic blood pressure (mm Hg) diastolic blood pressure (mmHg)
inflammation marker (blood) | change from baseline after 2 weeks
  high-sensitive c-reactive protein (mg/dl)
homocysteine | change from baseline after 2 weeks
  homocysteine (µmol/l)
holotranscobalamine | change from baseline after 2 weeks
  holotranscobalamine (pmol/l)
glucose (fasting) | change from baseline after 2 weeks
  glucose (fasting) (mmol/l)
insulin (fasting) | change from baseline after 2 weeks
  insulin (fasting) (mU/l)
hemoglobin A1c (fasting) | change from baseline after 2 weeks
  hemoglobin A1c (fasting) (%)
malodialdehyde modified LDL cholesterol | change from baseline after 2 weeks
  malodialdehyde modified LDL cholesterol (U/l)
fatty acid distribution in plasma lipids | change from baseline after 2 weeks
  fatty acid distribution in plasma lipids in % FAME
aspartate transaminase | change from baseline after 2 weeks
  aspartate transaminase (ASAT) in µmol/l*s
alanine transaminase | change from baseline after 2 weeks
  alanine transaminase (ALAT) in µmol/l*s
gamma-glutamyltransferase | change from baseline after 2 weeks
  gamma-glutamyltransferase (gGT) in µmol/l*s
lactate dehydrogenase | change from baseline after 2 weeks
  lactate dehydrogenase (LDH) in µmol/l*s
cholinesterase | change from baseline after 2 weeks
  cholinesterase in µmol/l*s
kalium | change from baseline after 2 weeks
  kalium in mmol/l
calcium | change from baseline after 2 weeks
  calcium in mmol/l
transferrin | change from baseline after 2 weeks
  transferrin (g/l)
ferritin | change from baseline after 2 weeks
  ferritin (µg/l)
iron | change from baseline after 2 weeks
  iron (mg/dl)
vitamin A | change from baseline after 2 weeks
  vitamin A (mmol/l)
vitamin D | change from baseline after 2 weeks
  vitamin D (nmol/l)
vitamin E | change from baseline after 2 weeks
  vitamin E (µmol/l)
vitamin B1 | change from baseline after 2 weeks
  vitamin B1 (nmol/l)
vitamin B6 | change from baseline after 2 weeks
  vitamin B6 (nmol/l)
vitamin B12 | change from baseline after 2 weeks
  vitamin B12 (pmol/l)
folic acid | change from baseline after 2 weeks
  folic acid (µg/l)
vitamin B2 | change from baseline after 2 weeks
  vitamin B2 (µg/l)
vitamin C | change from baseline after 2 weeks
  vitamin C (mg/l)
vitamin H | change from baseline after 2 weeks
  vitamin H (ng/l)
iodine (24 h urine) | change from baseline after 2 weeks
  iodine (µmol/l)
selenium (24 h urine) | change from baseline after 2 weeks
  selenium (µmol/l)
copper (24 h urine) | change from baseline after 2 weeks
  copper (µmol/l)
zinc (24 h urine) | change from baseline after 2 weeks
  zinc (µmol/l)
manganese (24 h urine) | change from baseline after 2 weeks
  manganese (nmol/l)
natrium (24 h urine) | change from baseline after 2 weeks
  natrium (mmol/l)
magnesium (24 h urine) | change from baseline after 2 weeks
  magnesium (mmol/l)
creatinine (24 h urine) | change from baseline after 2 weeks
  creatinine (mmol/24 h)
albumine (24 h urine) | change from baseline after 2 weeks
  albumine (mg/l)
uric acid (24 h urine) | change from baseline after 2 weeks
  uric acid (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich Schiller University, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No